CLINICAL TRIAL: NCT06320041
Title: Efficacy and Safety of Oliceridine for Moderate to Severe Acute Pain After Orthopedic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-2024-028
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low dose oxelidine group (Experimental): Oxelidine fumarate (10ml, 20mg) + normal saline 190ml diluted to 200ml. PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.35mg (3.5ml), locking time was 6min, and load was 1.5mg
  Interventions: Drug: Low dose oxelidine group
- high dose oxelidine group (Experimental): Oxelidine fumarate (10ml, 20mg) + normal saline 190ml diluted to 200ml. PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.5mg (5ml), locking time was 6min, and load was 1.5mg
  Interventions: Drug: High dose oxelidine group
- hydromorphone group (Active Comparator): Hydromorphone (6ml, 12mg) + normal saline (194ml) diluted to 200ml. PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.3mg (5ml), locking time was 6min, and load was 1mg
  Interventions: Drug: Hydromorphone group

INTERVENTIONS:
Drug: Low dose oxelidine group — Analgesic dose
  Arms: low dose oxelidine group
Drug: High dose oxelidine group — Analgesic dose
  Arms: high dose oxelidine group
Drug: Hydromorphone group — Analgesic dose
  Arms: hydromorphone group

SUMMARY:
The goal of this clinical trial] is to further explore the effectiveness and safety of oxelidine in the treatment of moderate to severe acute pain after orthopedic surgery. The main question it aims to answer is: Pain management after orthopaedic surgery provides more effective and safe drug options, provides new options for clinical treatment, and provides a scientific basis for clinical practice.

Participants will be asked to pain score in the different time, treatments they'll be given and use optimal drug. Researchers will compare analgesic effect of oxelidine of different dose.

DETAILED DESCRIPTION:
Induction and maintenance of anesthesia were the same in all patients, performed by the same anesthesiologist. The study Coordinator (Dr. He Kin Nang) used the Central randomization System software to randomly assign high-dose oxelidine fumarate (group H), low-dose oxelidine fumarate (group L) and hydromorphone (group M) in a ratio of 1:1:1. The distribution was concealed using the same opaque envelopes, which were sealed and stored in a locked cabinet, without the knowledge of the anesthesiologist and the follow-up physician.

The drugs for the study were prepared by an independent nurse anesthesiologist according to a randomized outcome code, using the drug's configuration:

Group L: oxelidine fumarate (10ml, 20mg) + 190ml normal saline diluted to 200ml, PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.35mg (3.5ml), locking time was 6min, load was 1.5mg; Group H: oxelidine fumarate (10ml, 20mg) + 190ml normal saline diluted to 200ml, PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.5mg (i.e. 5ml), locking time was 6min, load was 1.5mg; Group M: hydromorphone (6ml, 12mg) + normal saline (194ml) diluted to 200ml. PCIA parameters were set as follows: background infusion rate was 0, self-controlled dosage was 0.3mg (5ml), locking time was 6min, and load was 1mg.

The PCIA pump starts from the withdrawal of the tracheal catheter. When the patient's pain Numerical Evaluation Scale score (NRS) is ≥5, the effective pressure of the PCIA pump can be increased for 1-3 times according to the actual pain sensation. If the pain is still not relieved, the intravenous injection of hydromorphone 0.5-1mg (or drugs that can directly have a conversion relationship with morphine) can be slowly injected. The PCIA pump is stopped 48 hours after surgery. If the patient still feels pain and the NRS score is ≥5, 5-10mg of hydromorphone can be slowly injected intravenously (or drugs that can directly have a conversion relationship with morphine). In both groups, 200mg celecoxib (400mg daily) was taken orally at 08:00 and 16:00 each day from the first day after surgery (the second day of the study) as a multimodal analgesic regimen until the patients stopped the drug after no pain discomfort. If the study drug or remedial analgesic is still insufficient, the patient's study drug therapy is discontinued and the usual analgesic therapy as determined by the clinician is adopted.

Main study indicators: Area under the curve (AUC NRS-R0-72) of pain scores at rest 0-72 hours after surgery in the three groups. Pain scores 0 hours after surgery were replaced by pain scores 15 minutes after extubation.

Secondary study measures: The total amount of opioid relief analgesics converted into morphine 0-72 hours after surgery in the three groups; Three groups first used PCIA as a compression time for remedial analgesia; The area under the curve (AUCRNS-R0-72) of pain scores during exercise in the three groups at 0-72 hours after surgery was replaced by the pain scores during cough 15 minutes after extubation. NRS scores of resting and exercise at different time points in the three groups within 72 hours after operation; Duration of initial relief analgesia; 0-24h dosage of relief analgesic drugs; 0-48 hours of relief analgesia; 0-48The total number of HPCA pump presses and effective presses; The proportion of subjects who did not use remedial analgesia from 0 to 48h; Subject and investigator analgesic satisfaction scores.

Safety assessment (follow-up up to day 3) : exposure, follow-up of adverse events (AEs), respiration-related adverse events (hypoxemia, respiratory depression, hypoventilation), upper respiratory tract reactions (nausea, vomiting), drowsiness or sedation, fever, constipation, dizziness, headache, pruritus, etc.

ELIGIBILITY:
Inclusion Criteria:

1. elective orthopedic surgery under general anesthesia.
2. The patient can communicate normally and has the correct expression of pain

Exclusion Criteria:

1. Patients with advanced tumor
2. Other acute and chronic pain conditions are present
3. Severely obese (30 kg/m2)
4. Pregnant or lactating women
5. Allergy to opioids
6. Sleep apnea syndrome
7. Long-term opioid treatment
8. Patients with mental and nervous system diseases, gastrointestinal obstruction, chronic obstructive pulmonary disease or pulmonary heart disease, cardiovascular disease
9. Abnormal liver function during screening
10. Abnormal renal function during screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score at rest 0-72 hours after surgery | 1 h (hour), 6 h,12 h,18 h,24 h,32 h,40 h,48 h,60 h,72 h (hours) after surgery
  Patients' pain scores at rest were recorded from 0-72 hours after surgery.

SECONDARY OUTCOMES:
The total amount of opioid after operation. | 72 hours after surgery
  The total amount of opioid relief analgesics was converted into morphine after operation.
PCIA as a remedial analgesic press time | during procedure (The moment to remove the PCIA pump.)
  Record the number of PCIA pump compressions (including the number of effective and ineffective compressions)

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ma, Study Chair — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No